CLINICAL TRIAL: NCT02147457
Title: Prematurity as Predictor of Children's Cardiovascular-renal Health (PREMATCH)
Brief Title: Prematurity as Predictor of Children's Cardiovascular-renal Health
Acronym: PREMATCH
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: PREMATCH
Record Dates: First submitted 2014-04-09; First posted 2014-05-26 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2015-11

CONDITIONS: Endothelial Dysfunction; Sublingual Capillary Glycocalyx and Density; Visual Disturbances and Blindness; Ventricular Dysfunction, Left; Renal Impairment
Keywords: Prematurity; Extremely low birth weight; Phenotyping
MeSH Terms: conditions — Blindness; Ventricular Dysfunction, Left; Renal Insufficiency; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine collection Blood collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ELBW (CASES): Extremely low birth weights, born in 2000-2005, birth weight below 1000 grams, who were initially admitted (2000-2005) at the Neonatal Intensive Care Unit, UZ Leuven Belgium and have been well characterized and documented in the postnatal period.
- CONTROLS: Survivors (CASES) (n = 140) will be matched with two healthy controls. One control will be matched to sex, birth year and residential area and will be suggested by the index patient (e.g. school friend, neighbor), the second control will be age and sex matched from the area of the field.

SUMMARY:
Extreme preterm birth interferes with the development of the cardiovascular system. Both macro- as well as microvasculature undergoes extensive, organ specific maturation. Under normal fetal conditions, microvascular growth drives renal development and continues until 34-36 weeks of gestational age, while retinal vascular growth continues until term age. Studies show that there is association between low birth weight and cardiovascular dysfunction. According to the Barker hypothesis, this is due to nutritional shortage. In extreme preterm birth cases, this growth restriction is observed in neonatal life.

In adult life, this suboptimal growth is associated with impaired renal and (micro)vascular function, hypertension, glucose intolerance and cardiovascular disease. According to the Brenner hypothesis, disrupted renal development results in hyperfiltration and hypertension, a process that subsequently promotes itself and leads to renal impairment. We will investigate macro- and microvasculature in different organs, including eye, kidney, heart and sublingual mucosa in former preterm infants, now aged 8-13 years old and age-matched controls.

The expectation is that the results of this project will identify risk factors for cardiovascular-renal disease in the adult life of former preterm infants compared to the controls, while further analysis on mediators in neonatal life of this cardiovascular-renal outcome may provide new information on perinatal risk factors.

DETAILED DESCRIPTION:
STATE OF THE ART The cardiovascular system (both macro- and microcirculation) undergoes extensive maturation throughout fetal, perinatal and pediatric life. Extreme preterm birth interferes with the normal development of the cardiovascular and microcirculatory systems. Disruption in vascular ontogenesis leads to abnormalities in the microvascular structure and circulation in various organs, such as retina (retinopathy of prematurity [O'Connor et al.]), kidney (abnormal glomerulogenesis [Sutherland et al.]) and glycocalyx in sublingual capillaries [Nieuwdorp et al.], among microvascular-driven disruptions observed in other organs (e.g. periventricular leukomalacia [Takashima et al.], bronchopulmonary dysplasia [Gien et al.]). Besides the well known retinopathy of prematurity, microvascular growth drives glomerulogenesis in the kidney and terminates after 34-36 weeks of gestational age under normal fetal conditions.

Perinatal (fetal or neonatal) growth restriction or preterm birth therefore impairs glomerulogenesis [Sutherland et al., Abitbol et al., Barker et al., Faa et al., Gubhaju et al., Zaffanello et al.]. Other cardiovascular abnormalities following from premature birth in later life include decreased heart rate variability [Rakow et al.], endothelial dysfunction [Norman et al.] and hypertension [Abitbol et al., Keijzer-Veen et al.].

Epidemiological observations further confirm that former preterm born infants are indeed at increased risk to develop cardiovascular disease and chronic kidney disease during adulthood [Brenner et al., Carmody et al., Vieux et al., Zandi-Nejad et al.]. The concept that fetal and perinatal conditions affect normal cardiovascular and renal ontogeny is in itself not new. Epidemiological studies showed that there is an association between low birth weight and vascular dysfunction in later life, suggesting that vascular impairment in early life is a harbinger of a poorer long-term prognosis [Sutherland et al., Bacchetta et al., Keijzer-Veen et al., Puddu et al.]. Intra-uterine growth retardation and children small for gestational age can be regarded as a failure of a fetus to reach the genetic potential of growth due to nutritional deprivation, the so-called Barker hypothesis [Barker et al.]. In adult life, this early growth retardation is associated with impaired renal and (micro)vascular function, hypertension, glucose intolerance and cardiovascular disease [Sutherland et al., Abitbol et al., Faa et al., Zaffanello et al., Carmody et al., Keijzer-Veen et al.].

The same sequence of vascular impairment serving as an indicator for long-term prognosis applies to the (early) postnatal life of preterm infants. According to the Brenner hypothesis, the decreased number of nephrons causes hyperfiltration, sodium loss with activation of the renin-angiotensinaldosterone system and hypertension [Brenner et al.], a process that entails further nephron loss, predisposition to develop proteinuria and possibly chronic kidney disease [Vieux et al., Puddu et al.].

MOVING BEYOND THE CURRENT STATE OF THE ART This project aims to move beyond the state-of-the-art by studying association between macro- and microvascular structure and function in children (8-13 years) born prematurely (extremely low birth weights, ELBW, i.e. birth weight below 1000 grams), and sex- and age-matched controls. The specific strengths hereby are that this ELBW cohort has been well characterized on its perinatal aspects [George et al.]. The characterization in the postnatal period includes biometry, perinatal characteristics (e.g. Apgar score, drugs, respiratory support), creatinine trends in the first 6 weeks of postnatal life and psychomotor development (Bayley Scales of Infant Development) at the age of nine months and two years.

The phenotypes of interest for the current project include the micro- and macrocirculation, cardiac structure and function, endothelial function and renal anatomy and function during childhood. We hereby aim to apply state of the art methods (cf methodology section) to assess micro- and macrocirculatory function, combined with state of the art statistics and advanced tools (metabolomics, epigenetics) to explore epidemiological findings and its pathogenesis.

The expectation is that the results of this project will identify and quantify risk factors in former preterm infants for cardiovascular-renal disease when compared to control children, while we can also map early risk factors for cardiovascular-renal disease in adult life and pave the way for a better informed prevention of these complications. Finally, data collected in this specific cohort can be compared to data collected in other cohorts.

HYPOTHESIS We hypothesize that former ELBW infants, compared to controls following term birth, will be associated with changes in the macro- and microcirculation of the cardiovascular-renal system already in young children over and beyond what is currently known. These changes - even if subtle - are probably forerunners of cardiovascular-renal complications in adulthood. In addition, confounders (e.g. neonatal nutrition, neonatal treatment) documented in the early life may identify new approaches for early prevention.

OBJECTIVES Using a case-control design in a 1/2 proportion, this study aims to detect functional and structural changes in children after preterm birth (ELBW) compared with children born after normal gestation with normal weight. The phenotypic aspects considered cover micro- and macrovascular structures and function.

1. Endothelial function
2. Sublingual capillary glycocalyx and density
3. Retinal imaging and visual acuity
4. Left ventricular function
5. Renal anatomy and function
6. Structure and function of the carotid artery (intima-media thickness, distensibility, Young's elastic modulus), aortic pulse wave velocity and the systolic augmentation index.

MODULATORS Next, this project will search for host characteristics, life style and environmental factors (see below) that may further modulate the differences in youngsters born either prematurely (case, ELBW) and at term, as well as for circulating and urinary biomarkers that are associated with the observed differences, and may provide insight into the pathogenesis involved.

IDENTIFICATION OF PREDICTORS Based on the existing database of the early perinatal follow-up of the prematurely born infants, this project will attempt to construct models predicting increased risk of potentially clinically significant changes associated with preterm birth and vice versa (mediators in neonatal life may predict cardiovascular-renal outcome in adult life).

INTENTION TO LINK THESE DATASETS WITH OTHER COHORTS WITH SIMILAR OBSERVATIONS Finally, pooling of these cardiovascular phenotypic data in children with other cohorts, either or not former ELBW cases may provide opportunities for additional prediction model development, validation and subsequent secondary preventive strategies.

METHODOLOGY Methodology-related issues include phenotyping, database construction/quality control, modulators, predictors and statistics.

PHENOTYPING

1. Endothelial function will be assessed by 24h urinary microalbumin excretion and digital pulse wave amplitude hyperemic response (photoplethysmography,PPG). To determine amplitude changes of the digital pulse, the response of the PPG pulse wave amplitude to hyperemia will be calculated from the hyperemic fingertip as ratio of post-deflation PPG pulse to baseline amplitude (PAht/PAh0, PA=pulse amplitude, h=hyperemic finger, t=time interval, 0=baseline). To obtain this ratio, we will divide the PAht/PAh0 ratio by the corresponding ratio at the control hand (PAct/PAc0, c=control finger)[Kuznetsova et al.].
2. To measure sublingual capillary glycocalyx and density, videos (10 sec) of sublingual capillaries in 2 areas lateral of the frenulum and 3-4 cm anterior to the tongue base will be recorded, using orthogonal polarization spectral (OPS) and side stream dark field (SDF) imaging [Hubble et al.]. In our hands, the intra- and inter-observer reproducibility of capillary density is 10.2 and 13.4% respectively. The erythrocyte-endothelium gap is the gold standard for glycocalyx measurement in vivo [Nieuwdorp et al.], as endothelial glycocalyx allows limited access to erythrocytes. The perfused boundary region (PBR) hereby reflects glycocalyx thickness and integrity, increased PBR glycocalyx loss.
3. Retinal imaging will be performed using a Canon Cr-DGi (Canon Co Ltd, Kyoto, Japan) nonmydriatic retinal visualization system. After accommodation to darkness, 1 image/eye will be obtained [Liu et al.]. Trained observers will identify individual arterioles and venules, using a validated computer-assisted program IVAN (Vasculo-matic Nicola, Ophthalmology and Visual Science, University of Wisconsin-Madison[Sherry et al.]). In addition, we will investigate visual acuity (clearness of vision, spatial resolution of the visual processing system) by the non-invasive adapted Snellen charts without visual aids.
4. All children will undergo detailed assessment of left ventricular (LV) function through echocardiography. PREMATCH will hereby focus on early changes in diastolic and systolic LV function. In combination with tissue Doppler imaging (TDI), transmitral and pulmonary vein blood flows will be used to detect LV filling changes.
5. Renal anatomy and function will be assessed by 2-dimensional measurement, renal arterial Doppler blood flow measurement and 3-dimensional calculations. Creatinine clearance, 24h microalbuminuria and Cystatin C on peripheral blood (serum) will be quantified.
6. The structure and function of the carotid artery, aortic pulse wave velocity (PWV) and systolic augmentation index will be assessed as measures of macrovascular function and structure. We will use ultrasound to measure the local properties of the common carotid artery. diameter, distension, and intima-media thickness will be measured and averaged over 3 cardiac cycles in recordings consisting of >4 consecutive beats. Distensibility (103/kPa), compliance (mm²/kPa) and Young's elastic modulus will be calculated. Local application tonometry will be performed (SpyghmoCor system). Measurements will be performed at carotid, radial and femoral arteries. The local arterial pulse wave will be recorded as well as carotid-to-femoral and carotid-to-radial PWV (cf- and cr-PWV). The carotid and radial augmentation indexes will be measured directly at the carotid and radial arteries and the aortic augmentation index will be calculated from the radial signal by the validated generalized transfer function [Richart et al., Seidlerova et al., Mischak et al.].Furthermore, we will implement ambulatory assessment of central hemodynamics, using the Mobil-O-Graph 24h PWA Monitor (IEM GmbH, Stolberg, Germany), a validated monitor for 24h blood pressure monitoring, including the ARCSolver application, which allows pulse wave analysis of the central blood pressure and measuring of aortic PWV [Luzardo et al.].

DATABASE CONSTRUCTION/QUALITY CONTROL Trained nurses will code questionnaires, technicians will enter the data. For quality assurance, 10% of questionnaires will be randomly selected and recoded by another nurse. All data will be inputted twice by different technicians. Duplicate datasets will be compared with the PROC COMPARE application (SAS software) to trace input errors. Data coders and SAS programs will check for internal consistency of questionnaire replies. Non-Gaussian distributions will be normalized by proper transformation. As part of the quality control, descriptive statistics will be generated at 6 month intervals.

MODULATORS

* Anthropometric characteristics, by sex, age, height, weight, body mass index, span width, waist-tohip ratio, skinfolds (Harpenden Skinfold Caliper, Bedfordshire, UK).
* Matrix reasoning and spatial orientation tests (Wechsler), indicators of mental capability.
* Muscle strength, by grip strength.
* Sexual maturation, by Tanner scale.
* Office and self-measured home blood pressure, by Mobil-O-Graph 24h PWA monitor (IEM, Stolberg, Germany)
* Body composition, by Bodystat4000 (Bodystat Ltd, Douglas, UK)
* Questionnaire (education, medication use, habits, menarche (girls) and familial and personal history).
* Measurements on blood and 24h urine samples. Plasma, serum and urine samples will be divided into aliquots and stored (-20/-80°C) at the bio-bank of the Studies Coordinating Centre (SCC). Routine measurements include hemoglobin, hematocrit, red and white blood cell counts, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, differential white blood cells count, serum creatinine, uric acid, serum lipids (total, HDL-cholesterol), glycaemia and insulin. Measurements of metabolic, inflammatory and oxidative stress include: 8-hydroxy -2'-deoxyguanosine (8-OHdG), interleukin-6 and high sensitivity C-reactive protein[Pearson et al.]. Other measurements will be considered if enough samples are available (e.g. homeostasis model assessment index (HOMA)[Marcelis et al.], leptin, adiponectin [Marcelis et al., Yeon et al.], E-selectin, P-selectin, vascular adhesion molecule-1, plasma fibrinogen, tumor necrosis factor, superoxide dismutase or serum malondialdehyde[Rao et al., Sharma et al.]).

Measurements of 24h urine samples include volume, electrolytes, creatinine, micro-albumin, and aldosterone. Urinary proteomics will be done in collaboration with Prof Harald Mischak, SME Mosaiques (mosaiques-diagnostics.de) by capillary electrophoresis coupled to mass spectrometry according to standard operating procedures in an environment with proper quality control [Mischak et al.].

- GPS coordinates of residence. Meteorological data and data on airborne pollutants and fine particulate collected from the appropriate sources.

PREDICTORS In our published cohort [George et al.] on creatinemia in ELBW infants in the first 6 weeks of life, raised creatinemia reflected immaturity (e.g. gestational age, weight) and morbidity (Apgar, ventilation, retinopathy of prematurity, intraventricular hemmorrhage), but also treatment modalities (e.g. ibuprofen, steroids, parenteral nutrition). We will link the perinatal covariates and creatinine trends to the dataset of this study to explore to what extent perinatal data predict cardiovascular and renal outcome. Since also treatment modalities are included, this study will provide first data on long term cardiovascular and renal outcome following drug exposure.

ELIGIBILITY:
Inclusion Criteria:

* 151 cases are children who were initially admitted (2000-2005) at the Neonatal Intensive Care Unit, UZ Leuven Belgium as ELBW (birth weight below 1000 g) neonates and have been well characterized and documented in the postnatal period. Survivors (n = 140) will be matched with two controls.

Exclusion Criteria:

* If the control child is not in good health.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ELBW (birth weight below 1000 g) neonates and have been well characterized and documented in the postnatal period, survivors (n = 140) will be matched with two controls. One control will be matched to sex, birth year and residential area and will be suggested by the index patient, the second control will be age and sex matched from the area of the field center. All children considered are currently between 8 and 15 years of age.
  Based on GCP guidance and national law, parents or custodians will provide informed written consent, while the child has to provide informed assent.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function. | Baseline measurement. Cross-sectional study.
  Changes in the macro- and microcirculation of the cardiovascular-renal system:
  * Endothelial function
  * Sublingual capillary glycocalyx and density
  * Retinal imaging and visual acuity
  * Left ventricular function
  * Renal anatomy and function
  * Structure and function of the carotid artery (intima-media thickness, distensibility, Young's elastic modulus), aortic pulse wave velocity and the systolic augmentation index.

CONTACTS AND LOCATIONS:
Overall Officials: Karel M Allegaert, PhD, MD, Study Director — UZ Leuven, Belgium; Lotte Jacobs, PhD, Study Chair — UZ Leuven; Anke MJ Raaijmakers, MD, Principal Investigator — UZ Leuven, Belgium
Locations (1):
- Research Center, Eksel, Limburg, Belgium

REFERENCES:
- [Background] O'Connor AR, Stephenson T, Johnson A, Tobin MJ, Moseley MJ, Ratib S, Ng Y, Fielder AR. Long-term ophthalmic outcome of low birth weight children with and without retinopathy of prematurity. Pediatrics. 2002 Jan;109(1):12-8. doi: 10.1542/peds.109.1.12. PMID 11773536
- [Background] Sutherland MR, Gubhaju L, Moore L, Kent AL, Dahlstrom JE, Horne RS, Hoy WE, Bertram JF, Black MJ. Accelerated maturation and abnormal morphology in the preterm neonatal kidney. J Am Soc Nephrol. 2011 Jul;22(7):1365-74. doi: 10.1681/ASN.2010121266. Epub 2011 Jun 2. PMID 21636639
- [Background] Nieuwdorp M, Meuwese MC, Mooij HL, Ince C, Broekhuizen LN, Kastelein JJ, Stroes ES, Vink H. Measuring endothelial glycocalyx dimensions in humans: a potential novel tool to monitor vascular vulnerability. J Appl Physiol (1985). 2008 Mar;104(3):845-52. doi: 10.1152/japplphysiol.00440.2007. Epub 2007 Dec 27. PMID 18162484
- [Background] Takashima S, Itoh M, Oka A. A history of our understanding of cerebral vascular development and pathogenesis of perinatal brain damage over the past 30 years. Semin Pediatr Neurol. 2009 Dec;16(4):226-36. doi: 10.1016/j.spen.2009.09.004. PMID 19945657
- [Background] Gien J, Kinsella JP. Pathogenesis and treatment of bronchopulmonary dysplasia. Curr Opin Pediatr. 2011 Jun;23(3):305-13. doi: 10.1097/MOP.0b013e328346577f. PMID 21494147
- [Background] Abitbol CL, Rodriguez MM. The long-term renal and cardiovascular consequences of prematurity. Nat Rev Nephrol. 2012 Feb 28;8(5):265-74. doi: 10.1038/nrneph.2012.38. PMID 22371245
- [Background] Barker DJ. Fetal origins of coronary heart disease. BMJ. 1995 Jul 15;311(6998):171-4. doi: 10.1136/bmj.311.6998.171. PMID 7613432
- [Background] Faa G, Gerosa C, Fanni D, Nemolato S, Locci A, Cabras T, Marinelli V, Puddu M, Zaffanello M, Monga G, Fanos V. Marked interindividual variability in renal maturation of preterm infants: lessons from autopsy. J Matern Fetal Neonatal Med. 2010 Oct;23 Suppl 3:129-33. doi: 10.3109/14767058.2010.510646. PMID 20836739
- [Background] Gubhaju L, Sutherland MR, Black MJ. Preterm birth and the kidney: implications for long-term renal health. Reprod Sci. 2011 Apr;18(4):322-33. doi: 10.1177/1933719111401659. PMID 21427457
- [Background] Zaffanello M, Brugnara M, Bruno C, Franchi B, Talamini G, Guidi G, Cataldi L, Biban P, Mella R, Fanos V. Renal function and volume of infants born with a very low birth-weight: a preliminary cross-sectional study. Acta Paediatr. 2010 Aug;99(8):1192-8. doi: 10.1111/j.1651-2227.2010.01799.x. Epub 2010 Mar 14. PMID 20337778
- [Background] Rakow A, Katz-Salamon M, Ericson M, Edner A, Vanpee M. Decreased heart rate variability in children born with low birth weight. Pediatr Res. 2013 Sep;74(3):339-43. doi: 10.1038/pr.2013.97. Epub 2013 Jun 14. PMID 23770921
- [Background] Norman M, Martin H. Preterm birth attenuates association between low birth weight and endothelial dysfunction. Circulation. 2003 Aug 26;108(8):996-1001. doi: 10.1161/01.CIR.0000085069.09770.3D. Epub 2003 Aug 18. PMID 12925463
- [Background] Keijzer-Veen MG, Dulger A, Dekker FW, Nauta J, van der Heijden BJ. Very preterm birth is a risk factor for increased systolic blood pressure at a young adult age. Pediatr Nephrol. 2010 Mar;25(3):509-16. doi: 10.1007/s00467-009-1373-9. Epub 2009 Dec 15. PMID 20012998
- [Background] Brenner BM, Garcia DL, Anderson S. Glomeruli and blood pressure. Less of one, more the other? Am J Hypertens. 1988 Oct;1(4 Pt 1):335-47. doi: 10.1093/ajh/1.4.335. PMID 3063284
- [Background] Carmody JB, Charlton JR. Short-term gestation, long-term risk: prematurity and chronic kidney disease. Pediatrics. 2013 Jun;131(6):1168-79. doi: 10.1542/peds.2013-0009. Epub 2013 May 13. PMID 23669525
- [Background] Vieux R, Hascoet JM, Merdariu D, Fresson J, Guillemin F. Glomerular filtration rate reference values in very preterm infants. Pediatrics. 2010 May;125(5):e1186-92. doi: 10.1542/peds.2009-1426. Epub 2010 Apr 5. PMID 20368313
- [Background] Zandi-Nejad K, Luyckx VA, Brenner BM. Adult hypertension and kidney disease: the role of fetal programming. Hypertension. 2006 Mar;47(3):502-8. doi: 10.1161/01.HYP.0000198544.09909.1a. Epub 2006 Jan 16. PMID 16415374
- [Background] Bacchetta J, Harambat J, Dubourg L, Guy B, Liutkus A, Canterino I, Kassai B, Putet G, Cochat P. Both extrauterine and intrauterine growth restriction impair renal function in children born very preterm. Kidney Int. 2009 Aug;76(4):445-52. doi: 10.1038/ki.2009.201. Epub 2009 Jun 10. PMID 19516242
- [Background] Keijzer-Veen MG, Devos AS, Meradji M, Dekker FW, Nauta J, van der Heijden BJ. Reduced renal length and volume 20 years after very preterm birth. Pediatr Nephrol. 2010 Mar;25(3):499-507. doi: 10.1007/s00467-009-1371-y. Epub 2009 Dec 16. PMID 20013294
- [Background] Puddu M, Fanos V, Podda F, Zaffanello M. The kidney from prenatal to adult life: perinatal programming and reduction of number of nephrons during development. Am J Nephrol. 2009;30(2):162-70. doi: 10.1159/000211324. Epub 2009 Apr 2. PMID 19339773
- [Background] George I, Mekahli D, Rayyan M, Levtchenko E, Allegaert K. Postnatal trends in creatinemia and its covariates in extremely low birth weight (ELBW) neonates. Pediatr Nephrol. 2011 Oct;26(10):1843-9. doi: 10.1007/s00467-011-1883-0. Epub 2011 Apr 17. PMID 21499946
- [Background] Kuznetsova T, Szczesny G, Thijs L, Jozeau D, D'hooge J, Staessen JA. Assessment of peripheral vascular function with photoplethysmographic pulse amplitude. Artery Research. 2011;5(2):58-64.
- [Background] Hubble SM, Kyte HL, Gooding K, Shore AC. Variability in sublingual microvessel density and flow measurements in healthy volunteers. Microcirculation. 2009 Feb;16(2):183-91. doi: 10.1080/10739680802461935. PMID 19206003
- [Background] Liu Y-P, Richart T, Jin Y, Struijker-Boudierc HA, Staessen JA. Retinal arteriolar and venular phenotypes in a Flemish population: Reproducibility and correlates. Artery Research. 2011;5(2):72-9.
- [Background] Sherry LM, Wang JJ, Rochtchina E, Wong T, Klein R, Hubbard L, Mitchell P. Reliability of computer-assisted retinal vessel measurementin a population. Clin Exp Ophthalmol. 2002 Jun;30(3):179-82. doi: 10.1046/j.1442-9071.2002.00520.x. PMID 12010210
- [Background] Richart T, Thijs L, Nawrot T, Yu J, Kuznetsova T, Balkestein EJ, Struijker-Boudier HA, Staessen JA. The metabolic syndrome and carotid intima-media thickness in relation to the parathyroid hormone to 25-OH-D(3) ratio in a general population. Am J Hypertens. 2011 Jan;24(1):102-9. doi: 10.1038/ajh.2010.124. Epub 2010 Jul 1. PMID 20596035
- [Background] Seidlerova J, Bochud M, Staessen JA, Cwynar M, Dolejsova M, Kuznetsova T, Nawrot T, Olszanecka A, Stolarz K, Thijs L, Wojciechowska W, Struijker-Boudier HA, Kawecka-Jaszcz K, Elston RC, Fagard R, Filipovsky J; EPOGH investigators. Heritability and intrafamilial aggregation of arterial characteristics. J Hypertens. 2008 Apr;26(4):721-8. doi: 10.1097/HJH.0b013e3282f4d1e7. PMID 18327082
- [Background] Seidlerova J, Staessen JA, Nawrot T, Brand E, Brand-Herrmann SM, Casamassima N, Citterio L, Hasenkamp S, Kuznetsova T, Li Y, Manunta P, Richart T, Struijker-Boudier HA, Fagard R, Filipovsk Ygrave J. Arterial properties in relation to genetic variation in alpha-adducin and the renin-angiotensin system in a White population. J Hum Hypertens. 2009 Jan;23(1):55-64. doi: 10.1038/jhh.2008.113. Epub 2008 Sep 18. PMID 18800139
- [Background] Mischak H, Kolch W, Aivaliotis M, Bouyssie D, Court M, Dihazi H, Dihazi GH, Franke J, Garin J, Gonzalez de Peredo A, Iphofer A, Jansch L, Lacroix C, Makridakis M, Masselon C, Metzger J, Monsarrat B, Mrug M, Norling M, Novak J, Pich A, Pitt A, Bongcam-Rudloff E, Siwy J, Suzuki H, Thongboonkerd V, Wang LS, Zoidakis J, Zurbig P, Schanstra JP, Vlahou A. Comprehensive human urine standards for comparability and standardization in clinical proteome analysis. Proteomics Clin Appl. 2010 Apr;4(4):464-78. doi: 10.1002/prca.200900189. Epub 2010 Feb 3. PMID 21137064
- [Background] Pearson TA, Mensah GA, Alexander RW, Anderson JL, Cannon RO 3rd, Criqui M, Fadl YY, Fortmann SP, Hong Y, Myers GL, Rifai N, Smith SC Jr, Taubert K, Tracy RP, Vinicor F; Centers for Disease Control and Prevention; American Heart Association. Markers of inflammation and cardiovascular disease: application to clinical and public health practice: A statement for healthcare professionals from the Centers for Disease Control and Prevention and the American Heart Association. Circulation. 2003 Jan 28;107(3):499-511. doi: 10.1161/01.cir.0000052939.59093.45. No abstract available. PMID 12551878
- [Background] Marcelis M, Suckling J, Hofman P, Woodruff P, Bullmore E, van Os J. Evidence that brain tissue volumes are associated with HVA reactivity to metabolic stress in schizophrenia. Schizophr Res. 2006 Sep;86(1-3):45-53. doi: 10.1016/j.schres.2006.05.001. Epub 2006 Jun 27. PMID 16806836
- [Background] Yeon JY, Kim HS, Sung MK. Diets rich in fruits and vegetables suppress blood biomarkers of metabolic stress in overweight women. Prev Med. 2012 May;54 Suppl:S109-15. doi: 10.1016/j.ypmed.2011.12.026. Epub 2011 Dec 29. PMID 22226662
- [Background] Rao VS, Nagaraj RK, Hebbagodi S, Kadarinarasimhiah NB, Kakkar VV. Association of inflammatory and oxidative stress markers with metabolic syndrome in asian indians in India. Cardiol Res Pract. 2010 Dec 28;2011:295976. doi: 10.4061/2011/295976. PMID 21234321
- [Background] Sharma JB, Sharma A, Bahadur A, Vimala N, Satyam A, Mittal S. Oxidative stress markers and antioxidant levels in normal pregnancy and pre-eclampsia. Int J Gynaecol Obstet. 2006 Jul;94(1):23-7. doi: 10.1016/j.ijgo.2006.03.025. Epub 2006 May 30. PMID 16730727
- [Background] Luzardo L, Lujambio I, Sottolano M, da Rosa A, Thijs L, Noboa O, Staessen JA, Boggia J. 24-h ambulatory recording of aortic pulse wave velocity and central systolic augmentation: a feasibility study. Hypertens Res. 2012 Oct;35(10):980-7. doi: 10.1038/hr.2012.78. Epub 2012 May 24. PMID 22622282
- [Derived] Salaets T, Raaijmakers A, Zhang ZY, Yu YL, Wei DM, Staessen JA, Allegaert K. QTc intervals are not prolonged in former ELBW infants at pre-adolescent age. Pediatr Res. 2022 Sep;92(3):848-852. doi: 10.1038/s41390-021-01877-w. Epub 2021 Dec 2. PMID 34857877
- [Derived] Wei FF, Raaijmakers A, Melgarejo JD, Cauwenberghs N, Thijs L, Zhang ZY, Yu CG, Levtchenko E, Struijker-Boudier HAJ, Yang WY, Kuznetsova T, Kennedy S, Verhamme P, Allegaert K, Staessen JA. Retinal and Renal Microvasculature in Relation to Central Hemodynamics in 11-Year-Old Children Born Preterm or At Term. J Am Heart Assoc. 2020 Aug 4;9(15):e014305. doi: 10.1161/JAHA.119.014305. Epub 2020 Jul 31. PMID 32750311
- [Derived] Raaijmakers A, Zhang ZY, Levtchenko E, Simons SH, Cauwenberghs N, Heuvel LPVD, Jacobs L, Staessen JA, Allegaert K. Ibuprofen exposure in early neonatal life does not affect renal function in young adolescence. Arch Dis Child Fetal Neonatal Ed. 2018 Mar;103(2):F107-F111. doi: 10.1136/archdischild-2017-312922. Epub 2017 Jun 14. PMID 28615304
- [Derived] Raaijmakers A, Zhang ZY, Claessens J, Cauwenberghs N, van Tienoven TP, Wei FF, Jacobs L, Levtchenko E, Pauwels S, Kuznetsova T, Allegaert K, Staessen JA. Does Extremely Low Birth Weight Predispose to Low-Renin Hypertension? Hypertension. 2017 Mar;69(3):443-449. doi: 10.1161/HYPERTENSIONAHA.116.08643. Epub 2017 Jan 23. PMID 28115515